CLINICAL TRIAL: NCT01066598
Title: A Phase II Study of Rituximab Combined With Prednisone for the Initial Treatment of Chronic Graft Versus Host Disease
Brief Title: A Study of Rituximab Combined With Prednisone for the Initial Treatment of Chronic Graft Versus Host Disease (cGVHD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor Accrual
Sponsor: University Health Network, Toronto (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Dr. John Kuruvilla, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OZM-009 (GVHD-R01)
Record Dates: First submitted 2010-02-08; First posted 2010-02-10 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-08

CONDITIONS: Graft Versus Host Disease
Keywords: graft versus host disease; chronic graft versus host disease; cGVHD
MeSH Terms: conditions — Graft vs Host Disease; Bronchiolitis Obliterans Syndrome | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rituximab plus prednisone (Experimental): Rituximab 375 mg/m2 IV weekly X 4 doses + Prednisone 1 mg/kg/d Treat 61 Patients
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Rituximab 375 mg/m2 IV weekly X 4 doses + Prednisone 1 mg/kg/d
  Other Names: Rituxan

SUMMARY:
The purpose of this study is to determine the efficacy of the combination of rituximab and prednisone as initial therapy for chronic graft-versus-host disease (C-GVHD).

DETAILED DESCRIPTION:
Host antigen-presenting cells (APC) have an important role in the pathogenesis of chronic graft-versus-host disease (C-GVHD). B cell antigen-presenting cells may also be important in activating T cells in vivo. In a murine leukemia model, B cells have been shown to be important APCs in T cell responses. Rates of C-GVHD were shown to lower in a B cell deficient murine model when compared to mice that received rabbit immunoglobulin, and the rate of C-GVHD was even lower if grafts were depleted of B cells. It would appear that B cells have an important role as APCs in the pathogenesis of C-GVHD.

The chimeric anti-CD20 antibody Rituximab has been demonstrated to have activity in steroid-refractory graft versus host disease in a few small retrospective studies. Previous evidence in indolent lymphoma has demonstrated that Rituximab is a potent B-cell depleting agent. These observations suggest that B-cell depletion in graft versus host disease may be an effective therapy. Rituximab is currently being evaluated in two separate phase II studies currently enrolling patients who have had an allogeneic stem cell transplant (allo-SCT) or have developed GVHD.

The Dana Farber BMT program has recently published a phase II study examining the safety and effectiveness of rituximab monotherapy in the setting of steroid-refractory GVHD. Rituximab was administered weekly at the standard dose of 375 mg/m2. The clinical response rate was 70% and responses were limited to patients with cutaneous and musculoskeletal manifestations of C-GVHD. Median corticosteroid doses improved from 40 mg/day to 10 mg/day. The BMT program at Stanford is enrolling patients in a phase II study examining the impact of 4 weekly doses of 375 mg/m2 of Rituximab given starting on day +56 following allo-SCT in patients with chronic lymphocytic leukemia (CLL) or mantle cell lymphoma (MCL) in an attempt to prevent the development of subsequent GVHD.

These two studies will provide important phase II data regarding the safety and efficacy of Rituximab in the prevention of GVHD and the treatment of steroid-refractory GVHD. Another area of interest would be the initial treatment of GVHD. Although there is no universally recognized standard of care, corticosteroids form the backbone of treatment for GVHD and are either given as single agents or part of a combination therapy strategy with Cyclosporine A (CsA), Tacrolimus (FK506) or mycophenolate mofetil (MMF).

We propose a phase II study of rituximab in combination with prednisone as primary therapy for C-GVHD.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated symptomatic classical C-GVHD (with prior allogeneic stem cell transplant) requiring systemic therapy (defined as per NIH Consensus: a)At least 3 sites of organ involvement or individual organ score of at least 2, b)Patients on agents for GVHD prophylaxis (such as therapeutic dose or tapering cyclosporine A or tacrolimus) or patients that have received therapy for acute GVHD prior to enrollment are eligible
* Patients must be 18 years of age or older
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Patients must be accessible for treatment and follow-up. Patients registered on this trial must be treated and followed at the participating centre. Investigators must assure themselves the patients registered on this trial will be available for complete documentation of the treatment, adverse events response assessment and follow-up.
* Patient must be willing and able to complete the GVHD questionnaire
* For patients that have been started on prednisone therapy for cGVHD but otherwise meet all of the eligibility criteria, registration into this trial must occur no later than 14 days from the start of prednisone therapy.

Exclusion Criteria

* Uncontrolled infection at the time of study enrollment
* Recurrent malignancy at the time of study enrollment
* Previous systemic therapy for C-GVHD, a)Patients on agents for GVHD prophylaxis (such as therapeutic dose or tapering cyclosporine A or tacrolimus) or patients that have received therapy for acute GVHD prior to enrollment are eligible. b)Patients who have been restarted on full doses of agents used for GVHD prophylaxis (ie. cyclosporine A or tacrolimus) after these have tapered or discontinued are not eligible
* Inability to tolerate prednisone (includes pre-existing myopathy, diabetes with poor glycemic control, uncontrolled hypertension or fluid retention) or rituximab
* Usage of additional concurrent agents which could treat C-GVHD (ie. chemotherapeutic agents - cyclophosphamide, methotrexate or other immunosuppressive agents). Patients may be continued on stable or tapering dose of GVHD prophylaxis agents such as cyclosporine or tacrolimus, but must be tapered off by first study treatment
* The administration of anticancer therapies or other investigational agents is not permitted. Use of hematopoietic colony stimulating factors to manage blood counts is allowed.
* Sexually active males and females of childbearing potential unwilling to practice contraception during the study. Patients of childbearing potential must be willing to use a reliable method of birth control (i.e. double barrier method).
* Women of childbearing potential with either a positive or no pregnancy test at baseline or lactating. Postmenopausal women must have been amenorrheic for at least 12 months or surgically sterile to be considered of non-childbearing potential.
* Patients with immune deficiency are at increased risk of lethal infections. Therefore, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions.
* Patients with active hepatitis B are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
The efficacy of the combination of rituximab and prednisone as initial therapy for C-GVHD, which is defined as discontinuation of immunosuppressive therapy at 12 months with resolution of reversible manifestations of C-GVHD | 12 months

SECONDARY OUTCOMES:
To determine the response rate to treatment, defined as complete response plus partial response (PR) for rituximab and prednisone | 3 years
To determine the rate of recurrent C-GVHD following initial therapy with rituximab and prednisone | 3 years
To determine the relapse rate of the underlying malignancy for which the allo-SCT was performed from time of study registration after treatment with rituximab and prednisone | 3 years
To determine the rate of infection requiring treatment with anti-bacterial, anti-fungal or anti-viral therapy from time of study registration after treatment with rituximab and prednisone | 3 years
To determine overall survival of treated patients from time of study registration to a maximum of 3 years following study registration for patients receiving rituximab and prednisone | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: John Kuruvilla, Principal Investigator — University Health Network, Toronto
Locations (3):
- Canada (3):
  - Alberta Health Sciences - Tom Baker Cancer Centre, Calgary, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Princess Maragaret Hospital, Toronto, Ontario